CLINICAL TRIAL: NCT03386409
Title: Impact of Firearm Safety Device Distribution on Firearm Exposure in the Households of Patients With Mental Health Complaints
Brief Title: Firearm Storage Device Distribution to Families of Children With Mental Health Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Neil Uspal, Assistant Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 00000009
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Mental Health Disorders; Suicide or Selfinflicted Injury by Firearms and Explosives
Keywords: Injury prevention
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: In the first phase of the study, all participants are assigned to an observational baseline group. Once the enrollment milestone is met, the second phase of the study will open. In this phase, participants all receive the intervention of safe firearm storage device distribution. Participants are randomized to either the free device group, or the low cost ($5) device group.
Who Masked: Participant
Masking Description: Participants are not informed about their group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline (No Intervention): Participants receive the standard of care recommendations for safe firearm storage device usage.
- Free Device (Experimental): Participants receive the standard of care recommendations for safe firearm storage device usage In addition, the study intervention is provision of a free safe firearm storage device (lock box, trigger lock and/or cable lock) for firearm storage at the time of enrollment.
  Interventions: Behavioral: Free safe firearm storage device distribution
- Low Cost Device (Experimental): Participants receive the standard of care recommendations for safe firearm storage device usage. In addition, the study intervention is the provision of a low cost ($5) firearm storage device (lock box, trigger lock and/or cable lock) for firearm storage at the time of enrollment.
  Interventions: Behavioral: Low cost safe firearm storage device

INTERVENTIONS:
Behavioral: Free safe firearm storage device distribution — Participants in the experimental phase of the study receive a safe firearm storage device at the time of study enrollment. They are randomized to receive a free device. Safe firearm storage devices include a California Department of Justice-approved lock box, trigger lock and/or cable lock.
  Arms: Free Device
Behavioral: Low cost safe firearm storage device — Participants in the experimental phase of the study receive a safe firearm storage device at the time of study enrollment. They are randomized to receive a low cost ($5) device. Safe firearm storage devices include a California Department of Justice-approved lock box, trigger lock and/or cable lock.
  Arms: Low Cost Device

SUMMARY:
This study aims to describe the baseline rate of safe firearm storage device use in the homes of pediatric patients with mental health complaints treated in the Emergency Department (ED) and/or inpatient psychiatric unit of an urban tertiary pediatric hospital.

Follow-up data will be collected to ascertain any change(s) in the rate of safe firearm storage device use after patients have been treated for a mental health complaint, which includes standardized recommendations for safe firearm storage practices. This study also involves an intervention to distribute safe firearm storage devices to families of pediatric mental health patients during their hospital visit, and assesses whether safe storage device distribution impacts reported future rate of firearm safety device use.

DETAILED DESCRIPTION:
Firearm injuries are a significant cause of morbidity and mortality for children and teens. Access to firearms has been associated with suicide completion in the pediatric mental health population. Current practice in our pediatric Emergency Department (ED) and inpatient psychiatric unit is to screen all mental health patients for firearm access, and to recommend safe firearm storage practices. However, there is no data on the baseline rate of safe firearm storage device use in the homes of these patients, or on the effectiveness of providing these recommendations during hospitalization.

This study has two phases, a baseline and an intervention. During the baseline phase, the research team will study whether there is an improvement in safe firearm storage device use in the homes of participants 7 or 30 days after safe storage practices are recommended during an ED or inpatient psychiatric visit. During the intervention phase, in addition to the standard recommendation of safe storage practices during the visit, the research team will distribute firearm safety storage devices such as a lock box, trigger lock, and and/or cable lock to families at the time of study enrollment. The investigators will study whether there is an improvement in safe firearm storage device use in the homes of intervention participants after 7 or 30 days compared to the usual care group.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-17 years, inclusive
* Evaluated in the Emergency Department or inpatient psychiatric unit for a primary mental health complaint
* Presence of a firearm in household where patient resides at least one day per week and/or will reside for at least one of the 7 days following enrollment
* Accompanied by a parent or legal guardian
* Parent or legal guardian is proficient in English
* Parent or legal guardian is 18 years of age or older

Exclusion Criteria:

* Patient is 18 years of age or older
* Patient is not evaluated for a mental health complaint in the Emergency Department or inpatient psychiatric unit
* The adult participant has previously enrolled in the intervention phase of the study.
* Patient is accompanied by a parent/legal guardian who has previously enrolled a different child in the intervention phase of the study
* Patient is not accompanied by a parent or legal guardian during their PMBU or ED visit
* Parent or legal guardian accompanying patient does not reside and/or does not anticipate residing in the household with patient for any of the 7 days following enrollment and no other adult household member is present to consent Note: Adult household members may only consent to participate in this study if a parent or legal guardian is also present to provide informed consent.

For adult household members only:

Inclusion Criteria:

* 18 years of age or older
* Lives in same household as patient at least one day per week
* Has primary or shared responsibility for at least one firearm stored in the household
* Proficient in English

Exclusion Criteria:

* Resides in household with patient less than one day per week, and/or does not anticipate residing in the household with patient for any of the 7 days following enrollment
* Is not responsible for firearm storage in the home

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 255 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change in the number of unsecured firearms stored in the household. | 7 and 30 days post-enrollment
  Comparison in the participant-reported number of unsecured firearms stored in their household at the time of enrollment, 7 days post-enrollment, and 30 days post-enrollment.

SECONDARY OUTCOMES:
Proportion of participants with all firearms safely secured | Baseline, 7 days and 30 days post-enrollment
  Description of participants with all firearms secured using "triple safe" storage methods: firearms stored in a locked location, unloaded, and with ammunition stored in a separate, locked location
Proportion of participants who report storing fewer firearms in their homes at follow-up | Baseline, 7 days and 30 days post-enrollment
  Description of participants who report storing fewer firearms in their homes during follow-up surveys compared to reported number of firearms at baseline
Proportion of participants who report using a firearm safety storage device at follow-up | Baseline, 7 days and 30 days post-enrollment
  Description of participants who report using any safe firearm storage device at follow-up, change in any safe firearm storage device use from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Neil Uspal, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No